CLINICAL TRIAL: NCT05754190
Title: Assessing Symptom and Mood Dynamics in Pain Using the Smartphone Application SOMA
Status: Recruiting | Type: Observational
Sponsor: Brown University (Other)
Responsible Party: Principal Investigator, Frederike Petzschner, Assistant Professor, Psychiatry and Human Behavior; Carney Institute for Brain Science, Brown University
Other Study IDs: 2022003301
Record Dates: First submitted 2023-02-08; First posted 2023-03-03 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Chronic Pain; Acute Pain; Post Operative Pain; Fibromyalgia, Primary; Fibromyalgia, Secondary; Fibromyalgia; Irritable Bowel Syndrome; Chronic Headache Disorder; Chronic Migraine; Chronic Pelvic Pain Syndrome; Temporomandibular Joint Disorders; Endometriosis-related Pain; Arthritis; Chronic Low-back Pain; Failed Back Surgery Syndrome; Post Herpetic Neuralgia; Neuropathic Pain; Painful Diabetic Neuropathy; Painful Bladder Syndrome; Trauma-related Wound; Trauma, Multiple; Chronic Pain Syndrome; Chronic Shoulder Pain
Keywords: digital health; e-health; smartphone application; chronic pain; acute pain; symptom tracking; experience sampling methodology; ecological momentary assessment; pain self-management
MeSH Terms: conditions — Chronic Pain; Acute Pain; Pain, Postoperative; Fibromyalgia; Irritable Bowel Syndrome; Temporomandibular Joint Disorders; Arthritis; Failed Back Surgery Syndrome; Neuralgia, Postherpetic; Neuralgia; Diabetic Neuropathies; Cystitis, Interstitial; Multiple Trauma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Healthy Controls: [general study + sub study] No history of chronic pain
  Interventions: Device: SOMA pain manager smartphone application
- Acute pain: [general study] Pain duration < 3 months
  Interventions: Device: SOMA pain manager smartphone application
- Chronic pain: [general study] Pain duration > 6 months
  [sub-study] diagnosis of chronic low back pain, failed back surgery syndrome, or fibromyalgia
  Interventions: Device: SOMA pain manager smartphone application

INTERVENTIONS:
Device: SOMA pain manager smartphone application — SOMA is a smartphone application developed for acute and chronic pain patients to track daily mood and pain symptoms and overall activity.

SUMMARY:
This study relies on the use of a smartphone application (SOMA) that the investigators developed for tracking daily mood, pain, and activity status in acute pain, chronic pain, and healthy controls over four months.The primary goal of the study is to use fluctuations in daily self-reported symptoms to identify computational predictors of acute-chronic pain transition, pain recovery, and/or chronic pain maintenance or flareups. The general study will include anyone with current acute or chronic pain, while a smaller sub-study will use a subset of patients from the chronic pain group who have been diagnosed with chronic low back pain, failed back surgery syndrome, or fibromyalgia. These sub-study participants will first take part in one in-person EEG testing session while completing simple interoception and reinforcement learning tasks and then begin daily use of the SOMA app. Electrophysiologic and behavioral data from the EEG testing session will be used to determine predictors of treatment response in the sub-study.

DETAILED DESCRIPTION:
The investigators aim to study the temporal dynamics of pain and links between self-reported pain, mood/emotion, and activities using the daily tracking app SOMA. The experience of pain fluctuates over time, specifically in patients who suffer from chronic pain and those who are transitioning from an acute to a chronic state. Emotions and mood directly influence the experience of pain and may contribute to its chronification. The investigators will use statistical and computational approaches to better understand the dynamics of these reported daily symptoms to identify computational predictors of transition from acute to chronic pain. Specifically, the investigators hypothesize that certain symptom clusters will co-occur in time and be linked to external life events (e.g. emotional and physical stress) and emotional states (e.g. worry). Statistical/computational analysis of pain dynamics could therefore identify indicators for change points in the transition from acute to chronic pain.

ELIGIBILITY:
INCLUSION CRITERIA [General study]

* Chronic pain group:

  * Age above 18
  * Access to a personal smartphone and a stable internet connection
  * Average pain intensity score of greater than 3 in the past week or
  * Average pain interference score of greater than 3 in the past week or
  * Average pain distress score of greater than 3 in the past week
  * Pain duration: greater than 6 months
* Acute pain group:

  * Age above 18
  * Access to a personal smartphone and a stable internet connection
  * Average pain intensity score of greater than 3 in the past week

    ○ or
  * Average pain interference score of greater than 3 in the past week

    ○ or
  * Average pain distress score of greater than 3 in the past week
  * Pain duration: less than 3 months
  * Pain cause: Due to recent surgery, injury, acute illness, or childbirth (within the past 3 months)
* Healthy control group:

  * Age above 18
  * Access to a personal smartphone and a stable internet connection
  * Average pain intensity score of less than 3 in the past week
  * Average pain interference score of less than 3 in the past week
  * Average pain distress score of less than 3 in the past week
  * No surgery, injury, acute illness, or childbirth (within the past 3 months)
* In person EEG testing [Sub-Study only]:

  * Same as in General App Study Above and additionally:
  * Current diagnosis of Fibromyalgia, Chronic Low Back Pain or Failed Back Surgery Syndrome OR
  * No current or prior history of chronic pain
  * If participant has chronic low back pain or failed back surgery syndrome: are they planning to have either a radio-frequency ablation, back surgery, or spinal cord stimulation implant in the next few months
  * If participant has chronic low back pain or failed back surgery syndrome: have they received insurance approval for the procedure?
  * Ok with EEC/ECG measures

EXCLUSION CRITERIA [General study]

* Chronic pain group:

  * recent injury or surgery unrelated to the pain in the past 3 months
  * difficulty participating for technical/logistical issues (e.g., no computer, incompatible smartphone, can't commit to 4 months study participation);
  * Not fluent in English (difficulty understanding questions)
  * Current primary or metastatic cancer (organic cause of pain)
* Acute pain group:

  * History of Chronic Pain (Pain lasting for more than 6 months)
  * difficulty participating for technical/logistical issues (e.g., no computer, incompatible smartphone, can't commit to 4 months study participation);
  * Not fluent in English (difficulty understanding questions)
  * Current primary or metastatic cancer (organic cause of pain)
* Healthy control group:

History of Chronic Pain (Pain lasting for more than 6 months)

* difficulty participating for technical/logistical issues (e.g., no computer, incompatible smartphone, can't commit to 4 months study participation);
* Not fluent in English (difficulty understanding questions)

  -In person EEG testing [Sub-study only]: [will interfere with EEG data collection safety or quality]:
* Same as in General App Study Above and additionally:
* Baldness
* Pregnancy
* Dreadlocks
* Left-handedness
* Use of a wheelchair
* Heart failure diagnosis
* Current or prior experience with acute psychosis or mania
* implanted pacemaker, neurostimulator or any other head or heart implants
* require a hearing aid to hear properly
* claustrophobia
* metal fragments in the body

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Any person who fits the eligibility criteria for acute pain, chronic pain, or healthy control groups will be eligible to participate in the general parent study. Healthy controls or participants who have a diagnosis of chronic low back pain, failed back surgery syndrom or fibromyalgia are eligible to participate in the in-person EEG sub-study.
  Participants will be recruited from around Rhode Island and surrounding regions via online ads, listserv announcements, local healthcare clinics, rehab and nursing facilities, word of mouth, social media, and targeted newspaper/magazine/public transportation advertisements. Chronic pain participants eligible for the in-person EEG testing will be recruited via these methods as well as targeted recruitment with physicians treating these patients.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2023-06-20 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
[General Study] Acute-Chronic Pain Transition Probability | T1 [4 months of daily app use]
  Test whether daily affect (incl. mood), pain, activities, and other factors measured by the SOMA app can predict transition from acute to chronic pain, pain recovery, or pain maintenance using mixed effects linear regression model-based analyses to predict long- term pain scores such as pain intensity, unpleasantness, and/or interference

SECONDARY OUTCOMES:
[General Study] Feasibility of long-term app use | T1 [4 months of daily app use]
  Percentage of Soma users in acute and chronic pain groups who engage with the app for 4 months
[General Study] App Engagement | T1 [4 months of daily app use]
  Evaluate user engagement based on number of completed daily ESM assessments per person in the acute and chronic pain groups over the 4 months of app use
[General Study] Pain Dynamics | T0 [Baseline], T1 [4 months of daily app use], T2 [4 months], T3 [8 months], T4 [12 months]
  Test whether variability in daily pain location, intensity, unpleasantness, and interference, and daily pain expectations and prediction errors in the SOMA app can predict long-term pain scores in cross sectional between-group and longitudinal within-subject model-based analyses
[General Study] Activity Dynamics | T0 [Baseline], T1 [4 months of daily app use], T2 [4 months], T3 [8 months], T4 [12 months]
  Test whether types or number of daily activities, the effect of activities on pain, and activity expectations for the next day can predict long-term pain scores in cross sectional and longitudinal model-based analyses.
[General Study] Pain Beliefs | T0 [Baseline], T2 [4 months], T3 [8 months], T4 [12 months]
  Test whether questionnaire scores related to pain beliefs and personal/health history at T0 can predict long-term pain scores in cross sectional between-group and longitudinal within-subject model-based analyses
[General study] Mood Dynamics | T0 [Baseline], T1 [4 months of daily app use], T2 [4 months], T3 [8 months], T4 [12 months]
  Test whether variability in daily mood ratings and mood prediction errors can predict long-term pain scores in cross sectional between-group and longitudinal within-subject model-based analyses.
[General Study] Association between mood, pain, and activity | T0 [Baseline], T1 [4 months of daily app use], T2 [4 months], T3 [8 months], T4 [12 months]
  Assess the effect of mood, pain, pain prediction errors and mood prediction errors on future activities in cross sectional between-group and longitudinal within-subject model based analyses.
[General Study] Mood homeostasis as measured by SOMA app mood screens | T0 [Baseline], T1 [4 months of daily app use], T2 [4 months], T3 [8 months], T4 [12 months]
  Assess mood homeostasis using SOMA mood screens in cross sectional between-group and longitudinal within-subject model based analyses.
[General Study] Effect of Treatments on pain and mood as measured by SOMA app screens | T0 [Baseline], T1 [4 months of daily app use], T2 [4 months], T3 [8 months], T4 [12 months]
  Assess the effect of pain treatments on mood, pain and activities using the dedicated SOMA screens for these measures in cross sectional between-group and longitudinal within-subject model based analyses.
[General Study] Avoidance Learning task-computer game | T0 [Baseline], T2 [4 months]
  Test harm avoidance learning and generalization differences between pain patients and healthy controls using a computerized reinforcement learning game.
[Sub-Study] Avoidance Learning Task-EEG | T0 [Baseline]
  Test whether EEG frontal theta band power is increased during prediction error processing and harm avoidance contexts in a reinforcement learning task in cross-sectional between-group analyses.
[Sub-Study] Cardiac Interoceptive Attention Task-EEG | T0 [Baseline], T1 [4 months of daily app use], T2 [4 months], T3 [8 months], T4 [12 months]
  Test whether cross-sectional differences in EEG-measured Heartbeat-evoked potential (HEP) amplitude when attending to interoceptive vs exteroceptive stimuli differ between pain patients and healthy controls and test relationship to questionnaire measures at baseline and follow-up.
[Sub-study] Resting state- EEG | T0 [Baseline], T1 [4 months of daily app use], T2 [4 months], T3 [8 months], T4 [12 months]
  Test cross-sectional differences in EEG-measured Resting State Activity between pain groups and healthy controls and test relationships between resting EEG measures and questionnaire results at baseline and follow-up
[Sub-study] Treatment outcome prediction in chronic low back pain and failed back surgery syndrome patients | T0 [Baseline], T1 [4 months of daily app use], T2 [4 months], T3 [8 months], T4 [12 months]
  Test whether baseline EEG HEP and questionnaire measures predict pain scores at T3 following invasive back treatments (eg back surgery, spinal cord stimulation, radio-frequency ablation) that occur during T1.

CONTACTS AND LOCATIONS:
Overall Officials: Frederike H Petzschner, PhD, Principal Investigator — Brown University
Locations (1):
- Brown University, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No
Anyone interested in IPD should reach out to the Principal Investigator

REFERENCES:
- [Background] Voscopoulos C, Lema M. When does acute pain become chronic? Br J Anaesth. 2010 Dec;105 Suppl 1:i69-85. doi: 10.1093/bja/aeq323. PMID 21148657
- [Background] Apkarian AV, Baliki MN, Farmer MA. Predicting transition to chronic pain. Curr Opin Neurol. 2013 Aug;26(4):360-7. doi: 10.1097/WCO.0b013e32836336ad. PMID 23823463
- [Background] Baliki MN, Petre B, Torbey S, Herrmann KM, Huang L, Schnitzer TJ, Fields HL, Apkarian AV. Corticostriatal functional connectivity predicts transition to chronic back pain. Nat Neurosci. 2012 Jul 1;15(8):1117-9. doi: 10.1038/nn.3153. PMID 22751038
- [Background] Hashmi JA, Baliki MN, Huang L, Baria AT, Torbey S, Hermann KM, Schnitzer TJ, Apkarian AV. Shape shifting pain: chronification of back pain shifts brain representation from nociceptive to emotional circuits. Brain. 2013 Sep;136(Pt 9):2751-68. doi: 10.1093/brain/awt211. PMID 23983029
- [Background] Pincus T, Burton AK, Vogel S, Field AP. A systematic review of psychological factors as predictors of chronicity/disability in prospective cohorts of low back pain. Spine (Phila Pa 1976). 2002 Mar 1;27(5):E109-20. doi: 10.1097/00007632-200203010-00017. PMID 11880847
- See also: To find out more information about Petzschner lab research — https://fpetzschner.com/lab/
- See also: To find out more about how to download and use the SOMA Pain Manager app — https://somatheapp.com